CLINICAL TRIAL: NCT05254600
Title: A Randomized Controlled Trial of RISE for Nurse Leaders
Brief Title: RISE RCT for Nurse Leaders
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1839775
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Stress; Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will attend the RISE for Nurse Leaders program, which consists of nine 90-minute weekly psychoeducational group sessions facilitated by a licensed mental health counselor (LMHC)
  Interventions: Behavioral: RISE for Nurse Leaders Program
- Wait-list control group (Active Comparator): Control group will attend the RISE for Nurse Leaders program after the 3-month wait-list period
  Interventions: Behavioral: RISE for Nurse Leaders Program

INTERVENTIONS:
Behavioral: RISE for Nurse Leaders Program — Psychoeducational sessions designed to impact resilience, insight, self-compassion, and empowerment

SUMMARY:
The purpose of this study is to determine whether RISE for Nurse Leaders has a significant impact on nurse leaders' post-traumatic growth, resilience, insight, self-compassion, and empowerment, as well as mental well-being, in their personal lives and their working environment.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Licensed as an RN
* Unit-based nurse leader (i.e., assistant nurse manager, nurse manager) employed by AdventHealth in a hospital-based setting at the Altamonte Springs, Apopka, Celebration, Daytona Beach, DeLand, East Orlando, Fish Memorial, Kissimmee, New Smyrna Beach, Orlando, Palm Coast, Waterman, or Winter Park campus
* Able to speak, read, and understand English fluently
* Able to provide informed consent
* Willing and able to comply with all study procedures and requirements for the duration of the study.

Exclusion Criteria:

* Employed as a direct care nurse or in another level of nursing leadership (i.e., director of nursing, executive leader)
* A study participant of IRBNet #1504917 titled A Pilot Study of RISE for Nurse Managers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Growth Inventory | Group comparison from baseline to 3-month follow-up
  21 item questionnaire with a scale of 0-5, with 0 meaning I did not experience this change as a result of my crisis; and 5 meaning I experienced this change to a very great degree as a result of my crisis

SECONDARY OUTCOMES:
Brief Index of Affective Job Satisfaction | Group comparison from baseline to 3-month follow-up
  4 item questionnaire with a scale of 1-5, with 1 meaning strongly disagree; and 5 meaning strongly agree
Brief Resilience Scale | Group comparison from baseline to 3-month follow-up
  6 item questionnaire with a scale of 1-5, with 1 meaning strongly disagree; and 5 meaning strongly agree
General Self-Efficacy Scale | Group comparison from baseline to 3-month follow-up
  10 item questionnaire with a scale of 1-4, with 1 meaning not at all true; and 4 meaning exactly true
Perceived Stress Scale | Group comparison from baseline to 3-month follow-up
  10 item questionnaire with a scale of 0-4, with 0 meaning never; and 4 meaning very often
Professional Quality of Life (ProQOL) Scale | Group comparison from baseline to 3-month follow-up
  30 item questionnaire with a scale of 1-5 with 1 meaning never; and 5 meaning very often
Psychological Empowerment Instrument | Group comparison from baseline to 3-month follow-up
  12 item questionnaire with a scale of A-G, with A meaning very strongly disagree; and G meaning very strongly agree
Self-Reflection and Insight Scale | Group comparison from baseline to 3-month follow-up
  20 item questionnaire with a scale of 1-6; with 1 meaning strongly disagree; and 6 meaning strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy Scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. (pp. 35-37). Windsor, UK: NFER-NELSON
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kath LM, Stichler JF, Ehrhart MG. Moderators of the negative outcomes of nurse manager stress. J Nurs Adm. 2012 Apr;42(4):215-21. doi: 10.1097/NNA.0b013e31824ccd25. PMID 22441404
- [Background] Kath LM, Stichler JF, Ehrhart MG, Sievers A. Predictors of nurse manager stress: a dominance analysis of potential work environment stressors. Int J Nurs Stud. 2013 Nov;50(11):1474-80. doi: 10.1016/j.ijnurstu.2013.02.011. Epub 2013 Mar 21. PMID 23522937
- [Background] Labrague LJ, McEnroe-Petitte DM, Leocadio MC, Van Bogaert P, Cummings GG. Stress and ways of coping among nurse managers: An integrative review. J Clin Nurs. 2018 Apr;27(7-8):1346-1359. doi: 10.1111/jocn.14165. Epub 2018 Jan 24. PMID 29148110
- [Background] Lee H, Cummings GG. Factors influencing job satisfaction of front line nurse managers: a systematic review. J Nurs Manag. 2008 Oct;16(7):768-83. doi: 10.1111/j.1365-2834.2008.00879.x. PMID 19017239
- [Background] • Grant AM, Franklin J, Langford P. The Self-Reflection and Insight Scale: A new measure of private self-consciousness. Social Behavior and Personality. 2002; 30(8): 821-836.
- [Background] • Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005; 4(4): 287-291.
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Shirey MR, McDaniel AM, Ebright PR, Fisher ML, Doebbeling BN. Understanding nurse manager stress and work complexity: factors that make a difference. J Nurs Adm. 2010 Feb;40(2):82-91. doi: 10.1097/NNA.0b013e3181cb9f88. PMID 20124961
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] • Spreitzer GM. Psychological empowerment in the workplace: Dimensions, measurement, and validation. Academy of Management Journal. 1995; 38(5):1442-1465.
- [Background] • Stamm, B. H. (2009). Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL). http://www.proqol.org.
- [Background] Steege LM, Pinekenstein BJ, Arsenault Knudsen E, Rainbow JG. Exploring nurse leader fatigue: a mixed methods study. J Nurs Manag. 2017 May;25(4):276-286. doi: 10.1111/jonm.12464. Epub 2017 Feb 27. PMID 28244184
- [Background] • Thompson ER & Phua FTT. A Brief Index of Affective Job Satisfaction. Group & Organization Management. 2012; 37(3): 275-307.
- [Background] Warshawsky NE, Havens DS. Nurse manager job satisfaction and intent to leave. Nurs Econ. 2014 Jan-Feb;32(1):32-9. PMID 24689156